CLINICAL TRIAL: NCT02009956
Title: POST MARKETING STUDY OF THE ELIXIR DESyne® NOVOLIMUS ELUTING CORONARY STENT SYSTEM AND THE DESyne® BD NOVOLIMUS ELUTING CORONARY STENT SYSTEM IN THE TREATMENT OF PATIENTS WITH DE NOVO NATIVE CORONARY ARTERY LESIONS
Brief Title: EXCELLA Post-Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elixir Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ELX-CL-1004
Record Dates: First submitted 2013-12-06; First posted 2013-12-12 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DESyne Novolimus Eluting CSS (Other): Enrollment of up to 50 patients with up to two de novo native coronary artery lesions measuring between 2.5 and 4.0 mm in diameter and </= 34 mm in length receiving the DESyne Novolimus Eluting CSS.
  Interventions: Device: Subjects receiving DESyne Novolimus Eluting CSS

INTERVENTIONS:
Device: Subjects receiving DESyne Novolimus Eluting CSS

SUMMARY:
To evaluate long-term safety and performance of the DESyne Novolimus Eluting Coronary Stent System and the DESyne BD Novolimus Eluting Coronary Stent System

DETAILED DESCRIPTION:
DESyne and DESyne BD are not currently approved for sale in the United States.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be ≥18 years of age.
* The patient must have angina pectoris as defined by the Canadian Cardiovascular Society Classification, documented silent ischemia, or a positive functional study.
* The patient has a planned intervention of up to two lesions each coverable by a single stent located in separate major epicardial territories. Each lesion/vessel must meet the following criteria:
* De novo lesion
* The target lesion reference site must be visually estimated to be ≥ 2.5 mm and ≤ 4.0 mm in diameter.
* The target vessel must be a major coronary artery or major branch with a visually estimated stenosis of ≥ 50% and <100%.
* The visually estimated target lesion length must be ≤ 34 mm (DESyne Novolimus Eluting CSS) (Arm A)*.
* The visually estimated target lesion length must be ≤ 34 mm (DESyne BD Novolimus Eluting CSS) (Arm B)*
* ≥ TIMI 1 coronary flow.

  *Subject to commercial availability of product sizes in the specific region/country.
* The patient must be an acceptable candidate for coronary artery bypass surgery.
* Female subjects of childbearing potential must have a negative pregnancy test within seven (7) days before the procedure and must agree to use a reliable method of contraception from the time of screening through 12 months after the index procedure.
* The patient and the patient's physician agree to the follow-up schedule.
* The patient or guardian who has been informed of the nature of the study agrees to its provisions and has provided written informed consent, approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, mTOR inhibitor class drugs, cobalt chromium alloy, methacrylate or polylactide polymer, or sensitivity to contrast which cannot be adequately premedicated.
* The patient is a female, intending to get pregnant within the next year.
* Target vessel(s) require a staged procedure post index hospitalization discharge through 9 months of this index procedure.
* There will be an untreated significant lesion of > 40% diameter stenosis remaining proximal or distal to the target site after the planned intervention.
* Previous placement of a stent within 10 mm of the target lesion.
* Total occlusion or TIMI 0 coronary flow in the target vessel.
* Restenosis lesion
* The proximal target vessel or target lesion is severely calcified by visual assessment.
* Aorto-ostial location, unprotected left main lesion location, or a lesion within 5 mm of the origin of the LAD or LCX.
* Lesion involvement of a significant side branch (branch diameter > 2 mm) that would be covered by stenting.
* High probability that treatment other than PTCA or stenting will be required for treatment of the same lesion.
* The patient has suffered a myocardial infarction within the past 72 hours and the CK or CK-MB has not returned to normal at the time of the index procedure.
* The patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
* The patient suffered a stroke, transient ischemic neurological attack (TIA) or significant gastrointestinal (GI) bleed within the past six months.
* The patient has renal insufficiency as determined by a creatinine of > 2.0 mg/dl.
* The target lesion, or the target vessel proximal to the target lesion, contains thrombus.
* Documented left ventricular ejection fraction of ≤ 25%.
* The patient is a recipient of a heart transplant.
* The patient has extensive peripheral vascular disease that precludes safe sheath insertion or extreme anti-coagulation.
* The patient has other medical illness (i.e., cancer or congestive heart failure) that may cause the patient to be non-compliant with the protocol, confound the data interpretation or is associated withlimited life expectancy (i.e., less than one year).
* The patient is simultaneously participating in another investigational device or drug study. Patient must have completed the primary follow-up phase of any previous study. Trials with extended follow-up phases of now commercially available products are not considered investigational studies. Patients may be enrolled one time only in this trial.
* Patients who are unable or unwilling to cooperate with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-02-26 (Actual); Primary Completion 2015-03-02 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Device-oriented Composite Endpoint (DoCE) | 1, 9, 12, and 24 months
  Device-oriented Composite Endpoint (DoCE) at 1, 9, 12, and 24 months. DoCE is defined as cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization.

CONTACTS AND LOCATIONS:
Locations (4):
- Krankenhaus der Barmherzigen Brüder, Trier, Germany
- Jordan (2):
  - Jordan Hospital, Amman
  - King Abdullah University Hospital, Irbid
- Santiago de Compostela University Hospital Complex, Santiago de Compostela, Spain